CLINICAL TRIAL: NCT02860949
Title: Multimodal Drug Infiltration in Total Knee Arthroplasty: Is Posterior Capsular Infiltration Worth the Risk? A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Multimodal Drug Infiltration in Total Knee Arthroplasty: Is Posterior Capsular Infiltration Worth the Risk?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Boontanapibul, Krit, M.D. (Individual)
Responsible Party: Principal Investigator, piya pinsornsak, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-OT-6-130/57
Record Dates: First submitted 2016-07-24; First posted 2016-08-10 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Local anesthetic infiltration; Posterior capsular infiltration; Multimodal anesthesia; Knee arthroplasty; Pain control; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Bupivacaine; Morphine; Epinephrine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAI with PCI (Experimental): Local anesthetic infiltration with posterior capsular injection (Drug inject at Anterior soft tissue, Medial gutter area, Lateral gutter area and Posterior capsular area)
  Interventions: Drug: 0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg mixed NSS up to 100 mL; Procedure: Drug injection at Anterior soft tissue (25 mL)+Medial gutter area (25 mL)+Lateral gutter area (25 mL)+Posterior capsular infiltration (25 mL)
- LAI without PCI (Active Comparator): Local anesthetic infiltration without posterior capsular injection (Drug inject at Anterior soft tissue, Medial gutter area and Lateral gutter area)
  Interventions: Drug: 0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg mixed NSS up to 100 mL; Procedure: Drug injection at Anterior soft tissue (34 mL)+Medial gutter area (33 mL)+Lateral gutter area (33 mL

INTERVENTIONS:
Drug: 0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg mixed NSS up to 100 mL
Procedure: Drug injection at Anterior soft tissue (25 mL)+Medial gutter area (25 mL)+Lateral gutter area (25 mL)+Posterior capsular infiltration (25 mL)
  Arms: LAI with PCI
Procedure: Drug injection at Anterior soft tissue (34 mL)+Medial gutter area (33 mL)+Lateral gutter area (33 mL
  Arms: LAI without PCI

SUMMARY:
Multimodal local anesthetic infiltration (LAI) provides effective pain control in patients undergoing total knee arthroplasty (TKA). Some surgeons avoid posterior capsular infiltration (PCI) for fear of damaging posterior neurovascular structures. Data are limited on the added benefits of PCI using different combinations of local anesthetic agents. Therefore, the investigator wanted to know the effectiveness of pain control in LAI with and without PCI.

Half of participants received LAI with PCI, while the other half received LAI without PCI during total knee arthroplasty.

DETAILED DESCRIPTION:
Analgesic agents were bupivacaine, morphine, ketorolac and epinephrine. All patients received spinal anesthesia and patient controlled analgesia (PCA) for 24 hours post surgery. The surgical technique and postoperative medication protocols were identical in both groups. The visual analogue scale (VAS) for pain during activity and at rest, and morphine consumption were recorded at 6, 12, 18 and 24 hours postoperatively. LAI-related side effects, blood loss, length of hospital stay, and VAS for satisfaction were monitored. The reviewer was blinded to treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary OA of the knee, aged less than 80 years old, and able to understand and comply with the study procedures.

Exclusion Criteria:

* Previous drug dependency
* Inability to undergo a spinal block
* Allergy to study drugs
* Renal insufficiency
* Abnormal liver function
* History of stroke
* History of coronary artery disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The visual analogue scale (VAS) for pain | 24 hours after the operation

SECONDARY OUTCOMES:
Morphine consumption from patient controlled analgesia (PCA) | 24 hours after the operation
The visual analogue scale (VAS) for satisfaction | 24 hours after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Piya Pinsornsak, MD, Principal Investigator — Faculty of Medicine, Thammasat university
Locations (1):
- Thammasat university hospital, Pathum Thani, Klongluang, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safa B, Gollish J, Haslam L, McCartney CJ. Comparing the effects of single shot sciatic nerve block versus posterior capsule local anesthetic infiltration on analgesia and functional outcome after total knee arthroplasty: a prospective, randomized, double-blinded, controlled trial. J Arthroplasty. 2014 Jun;29(6):1149-53. doi: 10.1016/j.arth.2013.11.020. Epub 2013 Dec 2. PMID 24559684
- [Result] Rasmussen S, Kramhoft MU, Sperling KP, Pedersen JH. Increased flexion and reduced hospital stay with continuous intraarticular morphine and ropivacaine after primary total knee replacement: open intervention study of efficacy and safety in 154 patients. Acta Orthop Scand. 2004 Oct;75(5):606-9. doi: 10.1080/00016470410001501. PMID 15513495
- [Result] Shoji H, Solomonow M, Yoshino S, D'Ambrosia R, Dabezies E. Factors affecting postoperative flexion in total knee arthroplasty. Orthopedics. 1990 Jun;13(6):643-9. doi: 10.3928/0147-7447-19900601-08. PMID 2367246
- [Result] Maheshwari AV, Blum YC, Shekhar L, Ranawat AS, Ranawat CS. Multimodal pain management after total hip and knee arthroplasty at the Ranawat Orthopaedic Center. Clin Orthop Relat Res. 2009 Jun;467(6):1418-23. doi: 10.1007/s11999-009-0728-7. Epub 2009 Feb 13. PMID 19214642
- [Result] Pettine KA, Wedel DJ, Cabanela ME, Weeks JL. The use of epidural bupivacaine following total knee arthroplasty. Orthop Rev. 1989 Aug;18(8):894-901. PMID 2771438
- [Result] Mahoney OM, Noble PC, Davidson J, Tullos HS. The effect of continuous epidural analgesia on postoperative pain, rehabilitation, and duration of hospitalization in total knee arthroplasty. Clin Orthop Relat Res. 1990 Nov;(260):30-7. PMID 1977542
- [Result] Cook P, Stevens J, Gaudron C. Comparing the effects of femoral nerve block versus femoral and sciatic nerve block on pain and opiate consumption after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):583-6. doi: 10.1016/s0883-5403(03)00198-0. PMID 12934209
- [Result] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Result] Liu SS, Zayas VM, Gordon MA, Beathe JC, Maalouf DB, Paroli L, Liguori GA, Ortiz J, Buschiazzo V, Ngeow J, Shetty T, Ya Deau JT. A prospective, randomized, controlled trial comparing ultrasound versus nerve stimulator guidance for interscalene block for ambulatory shoulder surgery for postoperative neurological symptoms. Anesth Analg. 2009 Jul;109(1):265-71. doi: 10.1213/ane.0b013e3181a3272c. PMID 19535720
- [Result] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Result] Ben-David B. Complications of regional anesthesia: an overview. Anesthesiol Clin North Am. 2002 Sep;20(3):665-667, ix. doi: 10.1016/s0889-8537(02)00003-2. PMID 12298311
- [Result] Adibatti M, V S. Study on variant anatomy of sciatic nerve. J Clin Diagn Res. 2014 Aug;8(8):AC07-9. doi: 10.7860/JCDR/2014/9116.4725. Epub 2014 Aug 20. PMID 25302181
- [Result] Vloka JD, Hadzic A, April E, Thys DM. The division of the sciatic nerve in the popliteal fossa: anatomical implications for popliteal nerve blockade. Anesth Analg. 2001 Jan;92(1):215-7. doi: 10.1097/00000539-200101000-00041. PMID 11133630
- [Result] Tsukada S, Wakui M, Hoshino A. Postoperative epidural analgesia compared with intraoperative periarticular injection for pain control following total knee arthroplasty under spinal anesthesia: a randomized controlled trial. J Bone Joint Surg Am. 2014 Sep 3;96(17):1433-8. doi: 10.2106/JBJS.M.01098. PMID 25187581
- [Result] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Result] Krenzel BA, Cook C, Martin GN, Vail TP, Attarian DE, Bolognesi MP. Posterior capsular injections of ropivacaine during total knee arthroplasty: a randomized, double-blind, placebo-controlled study. J Arthroplasty. 2009 Sep;24(6 Suppl):138-43. doi: 10.1016/j.arth.2009.03.014. Epub 2009 Jun 10. PMID 19520544